CLINICAL TRIAL: NCT06796686
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Priming Regimen of 426c.Mod.Core-C4b Followed by HxB2.WT.Core-C4b Boosts, Both Adjuvanted With 3M-052 AF + Alum, in Adult Participants Without HIV and in Overall Good Health
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of a Priming Regimen of 426c.Mod.Core-C4b Followed by HxB2.WT.Core-C4b Boosts, Both Adjuvanted With 3M-052 AF + Alum, in Adult Participants Without HIV and in Overall Good Health
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 320
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: HIV
Keywords: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — aluminum sulfate; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): One fractional dose of 426c.Mod.Core-C4b and two bolus doses of HxB2.WT.Core-C4b
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: HxB2.WT.Core-C4b; Biological: 3M-052-AF adjuvant; Other: Aluminum hydroxide suspension (Alum) adjuvant; Other: Diluent
- Group 2A (Active Comparator): One fractional dose and one bolus dose of 426c.Mod.Core-C4b two bolus doses of HxB2.WT.Core-C4b
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: HxB2.WT.Core-C4b; Biological: 3M-052-AF adjuvant; Other: Aluminum hydroxide suspension (Alum) adjuvant; Other: Diluent
- Group 2B (Active Comparator): One split dose and one bolus of 426c.Mod.Core-C4b and two bolus doses of HxB2.WT.Core-C4b
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: HxB2.WT.Core-C4b; Biological: 3M-052-AF adjuvant; Other: Aluminum hydroxide suspension (Alum) adjuvant; Other: Diluent

INTERVENTIONS:
Biological: 426c.Mod.Core-C4b — 426c.Mod.Core-C4b is supplied at a concentration of 2 mg/mL, 0.55 mL per vial.
Biological: HxB2.WT.Core-C4b — HxB2.WT.Core-C4b is supplied at a concentration of 1 mg/mL, 0.5 mL per vial
Biological: 3M-052-AF adjuvant — immune response modifier (IRM)
Other: Aluminum hydroxide suspension (Alum) adjuvant — Alhydrogel.
Other: Diluent — Tris-NaCl buffer

SUMMARY:
This is a partially randomized, open-label phase 1 study to evaluate the safety and immunogenicity of a priming regimen of 426c.Mod.Core-C4b adjuvanted with 3M-052 AF + Alum followed by boosts with HxB2.WT.Core-C4b adjuvanted with 3M-052 AF + Alum.

The primary hypothesis is that the boosting with HxB2.WT.Core-C4b adjuvanted with 3M-052 AF + Alum will further mature broadly neutralizing antibody (bnAb)-precursor B-cell lineages elicited by 426c.Mod.Core-C4b adjuvanted with 3M-052 AF + Alum.

426c.Mod.Core-C4b adjuvanted with 3M-052 AF + Alum has been tested in HVTN 301 previously, whereas the HxB2.WT.Core-C4b will be first-in-human (FIH).

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrates an understanding of the study and is able and willing to complete the informed consent process.
2. 18 to 55 years old, inclusive, on day of enrollment.
3. Available for clinic follow-up through the last clinic visit, willing to undergo leukapheresis, and willing to be contacted after the last study-product administration, including for potential participation in additional studies.
4. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 320 PSRT are required prior to enrollment into HVTN 320.
5. In good general health according to the clinical judgment of the site investigator.
6. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgment of the site investigator.
7. Agrees to discuss their potential for HIV acquisition and agrees to prevention counseling.
8. Hemoglobin (Hgb):

   * ≥11.0 g/dL for AFAB volunteers
   * ≥13.0 g/dL for cisgender AMAB volunteers or for volunteers who have been on masculinizing hormone therapy for more than 6 consecutive months
   * ≥12.0 g/dL for AMAB volunteers who have been on feminizing hormone therapy for more than 6 consecutive months
   * For volunteers who have been on gender-affirming hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth.
9. White blood cell (WBC) count = 2,500 to 12,000/mm3 (WBC over 12,000/mm3 is not exclusionary if further evaluation shows general good health and if PSRT approval is granted).
10. Platelets = 125,000 to 550,000/mm3.
11. Alanine aminotransferase (ALT) < 2.5 × upper limit of institutional reference range.
12. Serum creatinine ≤ 1.1 × upper limit of normal (ULN) based on the institutional normal range.
13. Corrected total serum calcium level of ≥ 8.5 mg/dL. "Corrected" includes measurement of serum albumin.
14. Systolic blood pressure of 90 to < 140 mmHg and diastolic blood pressure of 50 to < 90 mmHg at screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mmHg systolic and 90 mmHg diastolic. A single measurement ≥ 160 systolic mmHg or 100 mmHg diastolic during the current study evaluation is exclusionary.
15. Negative HIV test results by one of the following options:

    * US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA)
    * Chemiluminescent microparticle immunoassay (CMIA)
    * Two negative results on HIV rapid tests (one of which must be FDA-approved CMIA)
16. Negative for anti-hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
17. Negative for hepatitis B surface antigen (HBsAg).
18. For AFAB or intersex at birth volunteers who are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"):

    * Must agree to use effective means of contraception from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.
    * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.

    Note: Persons who are NOT of pregnancy potential due to total hysterectomy or bilateral oophorectomy (verified by medical records) or menopause (no menses for ≥1 year) are not required to undergo pregnancy testing.
19. AFAB or intersex at birth volunteers must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

1. Volunteer who is breastfeeding/chestfeeding or pregnant.
2. Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT approval.
3. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
4. Previous or current recipient of an investigational HIV vaccine (previous placebo/control recipients are not excluded).
5. Receipt of non-HIV investigational vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) Emergency Use Listing (EUL), or if outside the US, by the national Regulatory Authority (RA) authorizing this clinical trial.
6. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as glucocorticoid use, ≥ prednisone 10 mg/day within 3 months prior to enrollment.
7. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
8. Previous receipt of VRC01 mAb or other CD4bs mAbs.
9. Receipt of any of the following within 4 weeks prior to enrollment:

   * Live replicating vaccine
   * Any mRNA-based vaccine with FDA licensure, FDA EUA, or WHO EUL
   * ACAM2000 vaccine > 28 days prior with a vaccination scab still present.
10. Receipt of any vaccine that is not covered in exclusion criterion #9 within 14 days prior to enrollment. Please note this includes replication-incompetent vaccines such as the Jynneos vaccine for the prevention of mpox (formerly known as monkeypox) disease.
11. Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
12. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of more than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
13. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any related vaccine or component of the study-vaccine regimen (eg, imiquimod).
14. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
15. Idiopathic urticaria within the past year.
16. Bleeding disorder diagnosed by a clinician that would make study procedures a contraindication.
17. History of seizure(s) within the past 3 years. Also exclude if volunteer has used medications to prevent or treat seizure(s) at any time within the past 3 years.
18. Asplenia or functional asplenia.
19. Active duty and reserve US military personnel.
20. Any other chronic or clinically significant condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of the study participant, hinder their ability to participate in the study, or affect their immune responses to study products. Such conditions include but are not limited to clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgment of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
21. Asthma is excluded if the participant has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days per week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium- to high-dose inhaled corticosteroids (> 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
    * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
22. A participant with a history of a PIMMC, either active or remote. Not exclusionary: (1) remote history of Bell's palsy (> 2 years ago) not associated with other neurologic symptoms and (2) mild psoriasis or other mild, uncomplicated, localized or dermatologic condition that does not require ongoing systemic treatment.
23. History of allergy to local anesthetic (Novocaine, Lidocaine).
24. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous (IV) drug use or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Local Signs and Symptoms within 14 Days Post-Vaccination | Within 14 days of receiving study vaccine
Incidence of Systemic Reactogenicity Signs and Symptoms within 14 Days Post-Vaccination | Within 14 days of receiving study vaccine
Incidence of Serious Adverse Events Over 52 Weeks Post-Vaccination | throughout the study and for 52 weeks following any receipt of the study product
Incidence of Medically Attended Adverse Events Over 52 Weeks Post-Vaccination | throughout the study and for 52 weeks following any receipt of the study product
Incidence of Adverse Events of Special Interest Over 52 Weeks Post-Vaccination | throughout the study and for 52 weeks following any receipt of the study product
Incidence of Adverse Events Leading to Withdrawal or Discontinuation Over 52 Weeks Post-Vaccination | throughout the study and for 52 weeks following any receipt of the study product
Frequency of CD4-bs-specific B cells before and approximately 12 weeks after each HxB2.WT.Core-C4b boost | 12 weeks after each HxB2.WT.Core-C4b boost
  assessed by flow cytometry
Evolution of CD4-bs-Specific BCRs Before and 12 Weeks After Each HxB2.WT.Core-C4b Boost | 12 Weeks After Each HxB2.WT.Core-C4b Boost
  Assessed by VH/VL Sequencing of Sorted B Cells

SECONDARY OUTCOMES:
Response rate of serum antibodies at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
  will be assessed against a panel of autologous, precursor-sensitive, and heterologous viruses as measured by TZM-bl assay
Potency of serum antibodies at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
  will be assessed against a panel of autologous, precursor-sensitive, and heterologous viruses as measured by TZM-bl assay
Neutralizing breadth of serum antibodies at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
  will be assessed against a panel of autologous, precursor-sensitive, and heterologous viruses as measured by TZM-bl assay
Response rate of Env-specific serum IgG binding antibodies will be assessed at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
Magnitude of Env-specific serum IgG binding antibodies will be assessed at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
Epitope specificity of Env-specific serum IgG binding antibodies will be assessed at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
Breadth of Env-specific serum IgG binding antibodies will be assessed at 2 weeks after the final 426c.Mod.Core-C4b prime and 2 weeks after each HxB2.WT.Core-C4b boost | 2 weeks after each HxB2.WT.Core-C4b boost
Magnitude of binding of Env-specific IgG binding antibodies | 2 weeks after each HxB2.WT.Core-C4b boost
Epitope specificity of Env-specific IgG binding antibodies | 2 weeks after each HxB2.WT.Core-C4b boost
Breadth of Env-specific IgG binding antibodies | 2 weeks after each HxB2.WT.Core-C4b boost
Potency of neutralizing antibodies | 2 weeks after each HxB2.WT.Core-C4b boost
  as measured by TZM-bl assay
Breadth of neutralizing antibodies | 2 weeks after each HxB2.WT.Core-C4b boost
  as measured by TZM-bl assay
Response rate of Env-specific serum IgG binding antibodies | at week 6 (visit 3) and week 17 (visit 5)
Magnitude of Env-specific serum IgG binding antibodies | at week 6 (visit 3) and week 17 (visit 5)
Epitope specificity of Env-specific serum IgG binding antibodies | at week 6 (visit 3) and week 17 (visit 5)
Breadth of Env-specific serum IgG binding antibodies | at week 6 (visit 3) and week 17 (visit 5)
Response rate of neutralizing antibodies | at week 6 (visit 3) and week 17 (visit 5)
  as measured by TZM-bl assay
Potency of neutralizing antibodies | at week 6 (visit 3) and week 17 (visit 5)
  as measured by TZM-bl assay
Breadth of neutralizing antibodies | at week 6 (visit 3) and week 17 (visit 5)
  as measured by TZM-bl assay
Frequency of CD4-bs-specific B cells | at week 15 (visit 4, prior to vaccination 2) and week 27 (visit 6, prior to vaccination 3)
  as measured by flow cytometry
Evolution of CD4-bs-specific BCRs | at week 15 (visit 4, prior to vaccination 2)
  assessed by VH/VL sequencing of sorted B cells
Response rate of Env-specific serum IgG binding antibodies | at approximately 4 weeks post the first prime (visit 3) and week 17 (visit 5)
Magnitude of Env-specific serum IgG binding antibodies | at approximately 4 weeks post the first prime (visit 3) and week 17 (visit 5)
Epitope specificity of Env-specific serum IgG binding antibodies | at approximately 4 weeks post the first prime (visit 3) and week 17 (visit 5)
Breadth of Env-specific serum IgG binding antibodies | at approximately 4 weeks post the first prime (visit 3) and week 17 (visit 5)
Response rate of neutralizing antibodies | at approximately 4 weeks post the first prime (visit 3) week 17 (visit 5)
  as measured by TZM-bl assay
Potency of neutralizing antibodies | at approximately 4 weeks post the first prime (visit 3) week 17 (visit 5)
  as measured by TZM-bl assay
Breadth of neutralizing antibodies | at approximately 4 weeks post the first prime (visit 3) week 17 (visit 5)
  as measured by TZM-bl assay
Frequency of CD4-bs-specific B cells | at week 15 (visit 4, prior to vaccination 2) and week 27 (visit 6, prior to vaccination 3).
  as measured by flow cytometry
Response rate of Env-specific serum IgG binding antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
Magnitude of Env-specific serum IgG binding antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
Epitope specificity of Env-specific serum IgG binding antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
Breadth of Env-specific serum IgG binding antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
Response rate of neutralizing antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
  as measured by TZM-bl assay
Potency of neutralizing antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
  as measured by TZM-bl assay
Breadth of neutralizing antibodies | at approximately week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
  as measured by TZM-bl assay
Frequency of CD4-bs-specific B cells | at week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)
  as measured by flow cytometry
Evolution of CD4-bs-specific BCRs | at week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)]
  assessed by VH/VL sequencing of sorted B cells
Response rate of Env-specific serum IgG binding antibodies | at week 29 (visit 7), week 39 (visit 8, prior to vaccination 4), week 41 (visit 9), and week 51 (visit 10)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Research Center; Emory University, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia Physicians & Surgeons, New York, New York
  - NY Blood Center CRS, New York, New York

IPD SHARING:
Plan to Share IPD: No